CLINICAL TRIAL: NCT02393404
Title: Enhancing Neuromuscular Performance and Central Nervous System Plasticity Through Functional Movement-power Training to Improve Balance Strategies in Children With Developmental Coordination Disorder: A Randomised Controlled Trial
Brief Title: Functional Movement-power Training for Children With Developmental Coordination Disorder: A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27100614
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PT-FMT (Experimental): Functional movement-power training group
  Interventions: Other: PT-FMT
- FMT alone (Experimental): Functional movement training group
  Interventions: Other: FMT alone
- Control (No Intervention): No intervention control group

INTERVENTIONS:
Other: PT-FMT — Physiotherapeutic functional movement-power training
  Arms: PT-FMT
Other: FMT alone — Physiotherapeutic power training
  Arms: FMT alone

SUMMARY:
Objective: To compare the effectiveness of functional movement-power training (PT-FMT), functional movement training (FMT) alone and no intervention in improving balance strategies and performance among children with developmental coordination disorder (DCD).

Design: A randomised controlled clinical trial. Sample: 87 children with DCD. Interventions: 12 weeks of PT and FMT or FMT alone in the two intervention groups.

Major outcomes: Sensory organisation test - balance strategy and composite scores; Movement Assessment Battery for Children - total impairment score and balance subscore; hand-held dynamometer measurements of lower limb muscle strength and time to peak force.

DETAILED DESCRIPTION:
With the growing numbers of children with dyspraxia in Hong Kong, the focus of paediatric rehabilitation services has shifted from severe motor disorders (e.g., cerebral palsy) to relatively minor motor problems such as developmental coordination disorder (DCD). Evidence-based treatment strategies must be developed to suit this changing need. Children diagnosed with DCD are characterised by marked impairment in motor functions. Poor balance ability is a major concern because it may predispose children to falls and affect their motor skill development. At present, rehabilitation regimes for DCD-affected children use functional movement training (FMT) to induce neural plastic changes in the central nervous system (CNS) and thus enhance functional (balance) performance. Less emphasis is placed on treating the neuromuscular impairments that might also affect functional outcomes. Recently, the investigators research team discovered that slowed hamstring muscle force production, a neuromuscular deficit, may be one of the causes of poor balance strategies in children with DCD, but no effective treatment strategy has yet been examined. Power training (PT) has been found to be effective in increasing the speed of muscle force production and balance in adults through various neuromuscular mechanisms. In this study, the investigators intend to treat both the CNS and peripheral neuromuscular deficits in DCD-affected children. Therefore, the investigators will incorporate PT into a conventional FMT regime. The investigators hypothesise that balance strategies and functional performance in children with DCD will be improved most by treating both the CNS and neuromuscular deficits. This hypothesis will be supported by the finding that PT with FMT is superior to FMT alone in improving balance strategies and functional performance in children with DCD.

Objective: To compare the effectiveness of PT-FMT, FMT alone and no intervention in improving balance strategies and performance among children with DCD. Design: A randomised controlled clinical trial. Sample: 87 children with DCD. Interventions: 12 weeks of PT and FMT or FMT alone in the two intervention groups.

Major outcomes: Sensory organisation test - balance strategy and composite scores; Movement Assessment Battery for Children - total impairment score and balance subscore; hand-held dynamometer measurements of lower limb muscle strength and time to peak force.

Anticipated results and clinical significance: DCD-affected children who receive FMT together with PT will have the best balance performance outcomes. If the results are positive, this training programme could be readily transferrable to clinical practice. This could have positive socio-economic implications, such as shorter treatment periods and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. a formal diagnosis of DCD based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR)
2. a gross motor composite score ≤ 42 on the Bruininks-Oseretsky Test of Motor Proficiency
3. 6-10 years old
4. attending a mainstream school; and (5) no intellectual impairment.

Exclusion Criteria:

1. diagnosis of an emotional, neurological or other movement disorder
2. significant congenital, musculoskeletal or cardiopulmonary disorders that might affect motor performance
3. receiving active treatments including traditional Chinese medicine
4. disruptive behaviour
5. unable to follow instructions thoroughly.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes in sensory organisation test balance strategy | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)
Changes in sensory organisation test composite scores | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)

SECONDARY OUTCOMES:
Changes in Movement Assessment Battery for Children total impairment score | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)
Changes in Movement Assessment Battery for Children balance subscore | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)
Changes in hand-held dynamometer measurements of lower limb muscle strength | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)
Changes in hand-held dynamometer measurements of lower limb muscle time to peak force | Baseline (0 month), 3-month post-intervention (3 months), and 3-month follow-up (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley SM Fong, PT, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Pokfulam, Hong Kong

REFERENCES:
- [Derived] Fong SSM, Guo X, Cheng YTY, Liu KPY, Tsang WWN, Yam TTT, Chung LMY, Macfarlane DJ. A Novel Balance Training Program for Children With Developmental Coordination Disorder: A Randomized Controlled Trial. Medicine (Baltimore). 2016 Apr;95(16):e3492. doi: 10.1097/MD.0000000000003492. PMID 27100457